CLINICAL TRIAL: NCT03077841
Title: Optimizing Preventative Adjuvant Linac-Based Radiation: The OPAL Trial a Phase II/III Study of Hypofractionated Partial Breast Irradiation in Women With Early Stage Breast Cancer
Brief Title: Hypofractionated Partial Breast Irradiation in Treating Patients With Early Stage Breast Cancer
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI Requested
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1035; NCI-2017-00476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1035 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-03-06; First posted 2017-03-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Ductal Breast Carcinoma In Situ; Early-Stage Breast Carcinoma; Invasive Breast Carcinoma; Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (hypofractionated partial breast irradiation) (Experimental): Patients undergo hypofractionated partial breast irradiation daily for 5 days. Patients may then receive 3 additional boost fractions at the discretion of the doctor.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Partial Breast Irradiation; Other: Questionnaire Administration
- Arm II (hypofractionated partial breast irradiation) (Active Comparator): Patients undergo standard breast irradiation daily for 15 days. Patients may then receive 5 additional boost fractions at the discretion of the doctor.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Partial Breast Irradiation

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Partial Breast Irradiation — Undergo hypofractionated partial breast irradiation
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (hypofractionated partial breast irradiation)

SUMMARY:
This phase II trial studies how well hypofractionated partial breast irradiation works in treating patients with early stage breast cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Treating only the part of the breast where the cancer started may lead to fewer side effects than standard treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. The risk of grade 2 or higher toxicity occurring during radiation and through the 6 month post-radiation follow up visit in patients treated with Optimizing Preventative Adjuvant Linac-based Radiation (OPAL) regimen.

SECONDARY OBJECTIVES:

I. To measure patient-reported cosmetic outcome, functional status, and breast pain with the OPAL regimen at 6 months, one year, two years, three years, four years, and five years after completing the OPAL regimen.

II. To measure physician-reported and photographically-assessed cosmetic outcome at 6 months, one year, two years, three years, four years, and five years after completing the OPAL regimen and to compare this to the best performing arm of 2010-0559.

III. To determine the 5-year risk of pathologically-confirmed invasive and/or in situ ipsilateral breast tumor recurrence (IBTR) for patients with ductal breast carcinoma in situ (DCIS) and early invasive breast cancer.

IV. To determine the 5-year risk of any recurrence of breast cancer, disease-free survival, and overall survival.

V. To determine maximal late (within 5 years) toxicities using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0 scale.

VI. To establish the feasibility of conducting multi-center radiation therapy trials within the MD Anderson Network.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo hypofractionated partial breast irradiation daily for 5 days. Patients may then receive 3 additional boost fractions at the discretion of the doctor.

ARM II: Patients undergo standard breast irradiation daily for 15 days. Patients may then receive 5 additional boost fractions at the discretion of the doctor.

After completion of study treatment, patients are followed up at 6 months, and at 1.5, 3.5, and 5.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pathologically-confirmed invasive breast cancer or ductal carcinoma in situ
* Pathologic T stage of Tis, T1, or T2 with total size of tumor =< 3 cm (this size criteria applies to both pure DCIS and invasive tumors)
* For patients with invasive breast cancer, pathologic N stage of N0, N0 (i-), or N0 (i+); pathologic staging of the axilla is not required for patients with pure DCIS
* Treatment with breast conserving surgery
* Unifocal primary tumor based on imaging and clinical assessment; microscopic multifocality is allowed
* Final surgical margins negative defined as no tumor on ink; lobular carcinoma in situ involving the final surgical margin will be disregarded
* For invasive cancers, the tumor must be estrogen receptor positive (defined as 10% or greater expression of estrogen receptor)
* If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed at least one month prior to study registration and the patient must have no evidence of disease for this prior non-breast cancer
* Patients must be enrolled on the trial within 12 weeks of the later of two dates: the final breast conserving surgical procedure or administration of the last cycle of cytotoxic chemotherapy
* Final criteria for eligibility established after simulation: The tumor bed can be readily visualized on simulation computed tomography (CT) and is localized to one quadrant or region of the breast that is amenable to partial breast irradiation

Exclusion Criteria:

* Tumor invasion of the skin including dermis, chest wall, or pectoralis musculature
* Any evidence of nodal positivity beyond pathologic stage of pN0(i+)
* Systemic chemotherapy prior to final breast conserving surgery
* Patient is pregnant or nursing
* History of therapeutic irradiation to the breast, lower neck, mediastinum or other area in which there could potentially be overlap with the affected breast
* History of prior invasive or in situ cancer in either breast
* Current diagnosis of bilateral breast cancer
* History of lupus or scleroderma

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 928 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2027-11-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Risk of grade 2 or higher toxicity | At 6 months post radiation
  Will evaluate whether or not the risk of this outcome is higher than the risk of grade 2+ toxic events in the best performing arm of our prior clinical trial that evaluated dosing schedules of whole breast irradiation (2010-0559).

SECONDARY OUTCOMES:
Patient-reported cosmetic outcome | At 6 months, one year, two years, three years, four years, and five years after completing the optimizing preventative adjuvant linac-based radiation (OPAL) regimen
  Patient-reported cosmetic outcome, functional status, and breast pain will be measured using the Breast Cancer Treatment Outcomes Scale (BCTOS) and will be compared for the IMPORT Low versus OPAL regimens. Each outcome will be evaluated both as a continuous variable and as a dichotomous variable with a cutpoint of >= 2.5, indicating a moderate or greater average change in the treated breast compared to the untreated breast which serves as an internal control. Will use descriptive statistics to summarize patient-reported cosmetic outcome, functional status, and breast pain over time. Box plots and graphical measures will be used to display the distribution of these outcomes over time and by treatment arm. Will conduct linear mixed models to assess changes in patient-reported cosmetic outcome, functional status, and breast pain scores over time. A random intercept will be included to account for within-subject correlations.
Physician-reported and photographically-assessed cosmetic outcome | At 6 months, one year, two years, three years, four years, and five years after completing the OPAL regimen
  Physician-reported cosmetic outcome, functional status, and breast pain will be measured using the Breast Cancer Treatment Outcomes Scale (BCTOS) and will be compared for the IMPORT Low versus OPAL regimens. Each outcome will be evaluated both as a continuous variable and as a dichotomous variable with a cutpoint of >= 2.5, indicating a moderate or greater average change in the treated breast compared to the untreated breast which serves as an internal control. Will use descriptive statistics to summarize patient-reported cosmetic outcome, functional status, and breast pain over time. Box plots and graphical measures will be used to display the distribution of these outcomes over time and by treatment arm. Will conduct linear mixed models to assess changes in patient-reported cosmetic outcome, functional status, and breast pain scores over time. A random intercept will be included to account for within-subject correlations.
Risk of pathologically-confirmed invasive and/or ipsilateral breast tumor recurrence (IBTR) | At 5 years
  Will be estimated using Kaplan and Meier product-limit estimator and modeled with Cox proportional hazards regression. IBTR will be measured from the date of treatment initiation to the date of last evaluation or IBTR. The 5-year risk of IBTR and any recurrence will be estimated along with 95% confidence intervals. Differences in each of these outcomes by treatment arm will be assessed using the log-rank test. Cox proportional hazards regression and/or competing risks regression will be used if needed to account for imbalance among treatment arms with respect to risk factors for these outcomes.
Risk of any recurrence of breast cancer | At 5 years
  Will be estimated using Kaplan and Meier product-limit estimator and modeled with Cox proportional hazards regression. Recurrence-free survival will be measured from the date of radiation treatment initiation to the earliest date of last clinic visit, date of first recurrence, or date of death. Differences in each of these outcomes by treatment arm will be assessed using the log-rank test. Cox proportional hazards regression and/or competing risks regression will be used if needed to account for imbalance among treatment arms with respect to risk factors for these outcomes.
Disease free survival (DFS) | At 5 years
  Will be estimated using Kaplan and Meier product-limit estimator and modeled with Cox proportional hazards regression. DFS will be measured from date of treatment initiation to the earliest date of last clinic visit, date of progression, date of recurrence, date of metastasis, or date of death. Differences in each of these outcomes by treatment arm will be assessed using the log-rank test. Cox proportional hazards regression and/or competing risks regression will be used if needed to account for imbalance among treatment arms with respect to risk factors for these outcomes.
Overall survival | At 5 years
  Will be estimated using Kaplan and Meier product-limit estimator and modeled with Cox proportional hazards regression. OS will be measured from the date of treatment initiation to the earliest date of last contact or death. Differences in each of these outcomes by treatment arm will be assessed using the log-rank test. Cox proportional hazards regression and/or competing risks regression will be used if needed to account for imbalance among treatment arms with respect to risk factors for these outcomes.
Incidence of adverse events | Up to 5 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4. Differences in National Cancer Institute CTCAE and Subjective, Objective, Management, Analytic (SOMA) toxicity by treatment arm will be evaluated using chi-square test or Fisher's exact test, as appropriate.
Feasibility of conducting multi-center radiation therapy trials within the MD Anderson Network | 5 years
  The trial will be considered feasible if >= 90% of enrolled and treated patients receive the prescribed radiation dosing per protocol without deviations.
TGF-beta analysis | Up to 5 years
  For this analysis, the primary outcome is grade 2 or higher breast fibrosis measured using the Subjective, Objective, Management, Analytic/Late Effects Normal Tissue Task Force scale at the 3.5 year follow up visit. The exposure of interest is the presence of at least one copy of the C-509T allele in germline deoxyribonucleic acid (DNA). Will also conduct exploratory analyses to assess the association of TGF-beta genotype with cosmetic outcome, other PROs, and toxicities. T-test or rank-sum test will be used for continuous measures and chi-squared or Fishers exact test will be used for categorical measures.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Smith, Principal Investigator — M.D. Anderson Cancer Center
Locations (15):
- United States (15):
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Community Cancer Center East, Indianapolis, Indiana
  - Covenant Medical Center Harrison, Saginaw, Michigan
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Saint Luke's Baptist Health System, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Reddy JP, Lei X, Bloom ES, Reed VK, Schlembach PJ, Arzu I, Mayo L, Chun SG, Ahmad NR, Stauder MC, Gopal R, Kaiser K, Fang P, Smith BD; OPAL Trial Investigators. Optimizing Preventive Adjuvant Linac-Based (OPAL) Radiation: A Phase 2 Trial of Daily Partial Breast Irradiation. Int J Radiat Oncol Biol Phys. 2023 Mar 1;115(3):629-644. doi: 10.1016/j.ijrobp.2022.09.083. Epub 2022 Oct 8. PMID 36216274

DOCUMENTS (1):
  • Informed Consent Form (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03077841/ICF_000.pdf